CLINICAL TRIAL: NCT06585865
Title: Resveratrol-mediated Changes in Extracellular Vesicle microRNA Cargo as a Novel Contributor to Resistance Training-induced Skeletal Muscle Adaptations in Older Adults
Brief Title: Strength Training and Resveratrol
Acronym: STaR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YI-2024-02; IRB 2024-587 (Other: Texas Tech University)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia; Anabolic Resistance
Keywords: Resistance training; Aging; Resveratrol; Sarcopenia; Extracellular Vesicles; MicroRNAs
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training; Resveratrol

STUDY DESIGN:
Intervention Model Description: After pre-testing, participants will be randomized to supplement with resveratrol (500 mg) or placebo for 14 weeks. All participants will complete two 6-week blocks of supervised strength training (full body, 3 days/week); each block will be followed by one week of testing.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (RSV) group (Experimental): Participants will be randomized to consume resveratrol (500 mg) daily for 14 weeks (two 6-week blocks of resistance training [supervised, full-body, 3 days/week] + one testing week [3 days] following each block) after the pre-testing period. Participants will be provided with 7 days' worth of supplements at a time in pre-filled pill boxes. Pill boxes will be refilled weekly and adherence monitored.
  Interventions: Behavioral: Resistance training; Dietary Supplement: Resveratrol 500 mg oral once daily.
- Placebo (Placebo Comparator): Participants will be randomized to consume placebo capsules (cellulose, visually identical to resveratrol capsules) daily for 14 weeks (two 6-week blocks of resistance training [supervised, full-body, 3 days/week] + one testing week [3 days] following each block) after the pre-testing period. Participants will be provided with 7 days' worth of supplements at a time in pre-filled pill boxes. Pill boxes will be refilled weekly and adherence monitored.
  Interventions: Behavioral: Resistance training; Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Resistance training — After pre-testing, participants will perform full-body strength training three times per week for two 6-week blocks. The acute program variables (sets, repetitions, training frequency) will follow a non-linear periodized, progressive design consisting of muti-joint and single-joint exercises. Exercise stress will be varied by using different exercises and loads. The two training blocks will be separated by a mid-intervention testing week, allowing for the study team to monitor participants' progress, communicate progress to participants to promote adherence, and adjust target loads as appropriate for the second half of the intervention. An additional testing week will follow the second 6-week block.
  Other Names: Strength training
Dietary Supplement: Resveratrol 500 mg oral once daily. — Participants will be randomized to consume resveratrol (500 mg) daily for 14 weeks (two 6-week blocks of resistance training [supervised, full-body, 3 days/week] + one testing week [3 days] following each block) after the pre-testing period. Participants will be provided with 7 days' worth of supplements at a time in pre-filled pill boxes. Pill boxes will be refilled weekly and adherence monitored.
  Arms: Resveratrol (RSV) group
Dietary Supplement: Placebo — Participants will be randomized to consume placebo capsules (cellulose, visually identical to resveratrol capsules) daily for 14 weeks (two 6-week blocks of resistance training [supervised, full-body, 3 days/week] + one testing week [3 days] following each block) after the pre-testing period. Participants will be provided with 7 days' worth of supplements at a time in pre-filled pill boxes. Pill boxes will be refilled weekly and adherence monitored.
  Arms: Placebo

SUMMARY:
The main goal of this study is to find out if supplementing with resveratrol improves skeletal muscle adaptations to strengthening exercise (resistance training or strength training) in adults age 60+, and to determine whether circulating vehicles of inter-organ communication (extracellular vesicles) and their cargo might help explain those responses. The investigators will also examine whether resveratrol supplementation improves blood vessel function and cognitive function (brain health) in response to strength training.

DETAILED DESCRIPTION:
After screening and providing informed consent, participants (healthy older adults, age 60+, minimally active) will be familiarized with the procedures and undergo pre-testing. After pre-testing, participants will be assigned to supplement with resveratrol or placebo (double-blinded) daily while undergoing a strength training intervention. Strength training will be performed 3x/week for two 6-week blocks, and each visit will be supervised by a member of the study team. An additional week of testing will follow each of the two 6-week blocks.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+
* Minimally active (less than 1 hour of structured exercise/week other than walking)
* No resistance training for the previous 6 months
* Not currently taking resveratrol supplements
* Stable medication, supplement, dietary, and physical activity regimens for the previous 3 months and no plans to change throughout the study period
* Body mass at least 110 lbs

Exclusion Criteria:

* Medical complications that could increase risk during exercise (e.g., cardiovascular disease, uncontrolled hypertension, type 1 or 2 diabetes, orthopedic contraindication to exercise, kidney disease, etc.)
* Cannabis or nicotine use
* Consume more than 7 alcohol-containing beverages per week

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Circulating extracellular vesicle microRNA profile | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Circulating extracellular vesicles will be isolated from plasma and their microRNA cargo will be sequenced.
Muscle torque | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Participants will be instructed to try and straighten their leg, against resistance, as forcefully as possible and maximal torque of the quadriceps assessed using a dynamometer.
Muscle fatigability | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Participants will perform 32 repetitions of knee extensions on a dynamometer and the change in torque from the beginning to the end will be used to indicate fatigability.
Muscle strength | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Participants will perform submaximal testing to assess strength on key exercises included in the strength training protocol.
Appendicular skeletal muscle mass index | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Assessed using dual-energy x-ray absorptiometry (DEXA)

SECONDARY OUTCOMES:
Waist-to-hip ratio | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Waist and hip circumferences measured using measuring tape
Vascular function | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Flow-mediated dilation
Cognitive function | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Grip strength | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Handgrip dynamometry
Lower body strength/endurance | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  Chair stand test (30 seconds)
Gait speed | During pre-, mid-, and post-testing (each separated by about 6 weeks)
  4-m walk test

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Levitt, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from human participants (other than large-scale data) will be deposited into the TTU Dataverse with restricted access - by request only. Data will be linked only with a unique code.
  MicroRNA sequencing data will be deposited to the Gene Expression Omnibus (GEO).
  The following will be submitted to accompany data:
  * Full study protocol
  * Names and descriptions of data sets
  * Annotated data collection forms
  * Data dictionary
  * Documentation of calculated variables
  * Any changes made to the protocol over time
  * Frozen datasets used for the primary publication, when applicable
Supporting Information: Study Protocol
Time Frame: Dr. Danielle Levitt (PI) will deposit data into the appropriate repositories. Data upload will occur when publications associated with each data set are submitted and made public (where applicable) upon acceptance.
Access Criteria: Human participants data (except large-scale data sets)- reasonable requests must be submitted to the TTU Dataverse.
  MicroRNA sequencing data will be available in large-scale output format with no identifiable information (unique code).